CLINICAL TRIAL: NCT04814030
Title: Transarterial Infusion of PD-1 Antibody Plus Chemoembolization and FOLFOX-based Chemtherapy for Unresectable BCLC C Stage HCC: a Single-arm, Phase 2 Clinical Trial
Brief Title: Transarterial Infusion of PD-1 Antibody Plus TACE-HAIC for Unresectable HCC: a Single-arm, Phase 2 Clinical Trial
Acronym: AIPD-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yunfei Yuan, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2021-060
Record Dates: First submitted 2021-03-23; First posted 2021-03-24 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: Trans hepatic arterial infusion of PD-1 antibody, chemoembolization and FOLFOX-based chemotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AIPD-1 (Experimental): Trans hepatic artery infusion of PD-1 antibody, chemoembolization, FOLFOX-based infusion chemotherapy
  Interventions: Drug: PD-1 inhibitor

INTERVENTIONS:
Drug: PD-1 inhibitor — Transarterial hepatic chemoembolization and FOLFOX-based infusion
  Other Names: TACE-HAIC

SUMMARY:
Hepatocellular carcinoma (HCC) is a common disease in East Asia. Less than 20% of newly diagnosed patients can undergo radical resection. For those with unresectable BCLC C stage, transarterial chemotherapy and targeted therapy are recommend to prolong survival. Recently, FOLFOX (Oxaliplatin and 5-fluorouracil) based hepatic artery infusion chemotherapy (HAIC) exhibited high response rate for unresectable HCC. Transartery infusion of agents provide promising outcome when compared systemic infusion. Furthermore, our pilot study showed TACE combined HAIC (TACE-HAIC) had better tumor response, with low progression disease rate. Whether TACE-HAIC plus hepatic artery infusion PD-1 antibody would improve survival for unresectalbe BCLC C stage patients is still unknown. A single arm, phase 2 clinical trial is aimed to answer this question.

ELIGIBILITY:
Inclusion Criteria:

* BCLC C stage with unresectable diseasehigh-recurrence risk factor;
* Child-Pugh A or B (7 score) liver function;
* Anticipated survival more than 3 moths

Exclusion Criteria:

* Pregnant woman or sucking period;
* With other malignant cancer;
* Received anti-HCC therapy before this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 12 month
  defined as the sum of complete responses (CRs) and partial responses (PRs) over a specified time period

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No